CLINICAL TRIAL: NCT02688400
Title: An International, Multicentre, Double-blind, Randomised Study of the Effect of Diacerein vs Celecoxib on Symptoms and Structural Changes in Symptomatic Knee Osteoarthritis Patients as Assessed by Magnetic Resonance Imaging
Brief Title: Effect of Diacerein vs Celecoxib on Symptoms and Structural Changes in Symptomatic Knee Osteoarthritis
Acronym: DISSCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TRB Chemedica International SA (Industry)
Collaborators: ArthroLab Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAR-INT-14-01; 2015-002933-23 (EudraCT Number)
Record Dates: First submitted 2016-02-10; First posted 2016-02-23 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Osteoarthritis, Knee; Diacerein; Celecoxib; Phase III; Phase IV; Phase III-IV; Canada; Spain; Austria; Czech Republic; WOMAC
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — diacerein; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diacerein (Experimental): One placebo capsule once daily in the morning (breakfast) and one diacerein 50 mg capsule once daily in the evening (dinner) for the first month, then diacerein capsules twice daily with meals in the morning (breakfast) and the evening (dinner).
  Interventions: Drug: Diacerein; Drug: Placebo
- Celecoxib (Active Comparator): One celecoxib 200 mg capsule once daily in the morning (breakfast) and one placebo capsule once daily in the evening (dinner).
  Interventions: Drug: Celecoxib; Drug: Placebo

INTERVENTIONS:
Drug: Diacerein
  Other Names: Artrodar, Artrodarin, Artrolyt, Fisiodar, Galaxdar, Glizolan, Verboril
  Arms: Diacerein
Drug: Celecoxib
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Placebo

SUMMARY:
Osteoarthritis (OA) of the knee is the most frequent cause of knee pain after the age of 50 years. OA is a joint disease characterised by articular cartilage loss associated with structural changes in the cartilage and adjacent structures. The main symptoms are pain and functional disability. The goals of OA therapy are to decrease pain and maintain or improve joint function. There is evidence that diacerein has both a symptomatic and a structural effect on cartilage, and clinical studies suggest that diacerein therapy significantly decreases OA symptoms when compared to placebo. Diacerein has been shown to inhibit interleukine-1 (IL-1β), and down-regulated IL-1β stimulated secretion of metalloproteinases and aggrecanases, and thereby prevent breakdown of cartilage by these enzymes. Diacerein has no effect on the synthesis of prostaglandins, and therefore no effect on the upper intestinal tract. The purpose of this phase III-IV international, multicentre, double-blind, non-inferiority, randomised, controlled study is to determine the efficacy and safety of diacerein vs. celecoxib on symptoms after 6 months of treatment, and on structural changes after 2 years of treatment in knee OA patients as assessed by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The study was a phase III (Canada and Belgium) or IV (Spain, Austria and Czech Republic) international, multicentre, double-blind, randomized, controlled, parallel-groups, symptom-modifying and structure-modifying clinical study of Diacerein (50 mg twice daily) versus Celecoxib (200 mg once daily).

It was planned that 400 patients (males and females) of at least 50 years of age would take part in the study (approximately 150 patients in Canada and 250 patients in European countries). All patients were included after a Screening Visit (washout of previous medication for osteoarthritis) and randomized at the Inclusion Visit (Day 0) in 2 treatment groups of 200 patients as follows:

* Diacerein arm: one 50 mg capsule taken once a day for one month and 50 mg twice daily thereafter (n = 200 patients),
* Celecoxib arm: one 200 mg capsule once daily (n = 200 patients). All patients were assessed at Screening Visit (Visit 1), Inclusion (Visit 2, Day 0), Visit 3 (Day 60), Visit 4 (Day 120) and Visit 5 (Day 182 / early termination) (symptom study).

The duration of the double-blind study for each patient was up to 182 ± 7 days for the symptom study.

During the study, patients were allowed to take acetaminophen 500 mg, to a maximum of 2 g per day, dispensed at each visit by the investigator for rescue therapy.

Pain and other functional symptoms were primary analysed after 6 months (182 days) of treatment (symptom study).

Acetaminophen was dispensed during the study as rescue therapy in case of pain. However, it was asked to discontinue acetaminophen 48 hours before each study procedure/assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of at least 50 years of age;
* Patients followed in an ambulatory clinic;
* Patients presenting primary OA of the knee according to American College or Rheumatology (ACR) criteria;
* Patients with OA of radiological stages 2 and 3 according to Kellgren-Lawrence;
* Patients with a minimum joint space width ≥ 2 mm in the medial tibio-femoral compartment on standing knee X-ray (MRI structural study only);
* Patients with knee pain on most days of the month before entering into the study;
* Patients with a VAS pain score (0-100 mm) while walking on a flat surface ≥ 40 mm (Visit 1 (Screening) and Visit 2 (Inclusion Visits));
* Patients with no clinically significant laboratory abnormalities in the judgment of the investigator;
* Female patients who are postmenopausal with confirmed amenorrhea for at least one year before entering this study and those who underwent tubal ligation, oophorectomy or hysterectomy must agree to a hormonal (folliculo-stimulating hormone [FSH]) dosage at Screening visit ;
* Patients agreeing to sign the Informed Consent Form prior to any study-related activities after having been clearly informed of its methods and constraints;
* Patients not taking part in another clinical study;
* Patients agreeing to respect the protocol by attending the visits related to the study.

Exclusion Criteria:

Criteria related to individual characteristics of the patient

* Patients with secondary knee OA;
* Patients with known hypersensitivity to Diacerein or to anthraquinone-containing product, hypersensitivity to Celecoxib, who have demonstrated allergic-type reactions to sulphonamides, experienced asthma, urticaria or allergic-type reactions after taking sulphonamides, aspirin (acetyl salicylic acid [ASA]), lactose, non-steroidal anti-inflammatory drugs [NSAIDs], acetaminophen or paracetamol;
* Patients with a known history of diarrhoea, more particularly if 65 years of age and older;
* Patients with active malignancy of any type or history of a malignancy within the last five years other than basal cell carcinoma;
* Patients with other bone and articular diseases (antecedents and/or current signs) such as; chondrocalcinosis, Paget's disease of the ipsilateral limb to the target knee, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis, seronegative spondylo-arthropathy, mixed connective tissue disease, collagen vascular disease, psoriasis, inflammatory bowel disease;
* Pain in other parts of the body greater than the knee pain that could interfere with the evaluation of the index joint;
* Patients with fibromyalgia;
* Patients with isolated knee lateral compartment OA defined by joint space loss in the lateral compartment only;
* Patients with Class IV functional capacity using the American Rheumatism Association criteria;
* Patients who have had surgery in any lower limb or arthroscopy, aspiration or lavage in any lower limb joint within 180 days of the Inclusion Visit (Visit 2);
* Patients who have had meniscal surgery on the study knee;
* Patients who have undergone total knee replacement in the contralateral knee within 180 days prior to the Screening Visit (Visit 1);
* Patients with co-morbid conditions or joint deformity that restrict knee function;
* Patients with a history of heart attack or stroke, or who have had serious diseases of the heart such as congestive heart failure (functional classes II-IV of the New York Heart Association [NYHA]);
* Patients who have significant risk factors for heart attack or stroke will be assessed carefully. Risk factors for heart attack and stroke include high blood pressure (treated or untreated), high cholesterol, diabetes and smoking. The global risk assessment will be assessed using the American Heart Association (AHA) assessment of cardiovascular (CV) risk tables. Patients with high risk of CV events, according to the tables, will be excluded;
* Patients with any significant diseases or conditions, including emotional or psychiatric disorders and substance abuse that, in the opinion of the Investigator, are likely to alter appreciation of OA symptoms or the patient's ability to complete the study;
* Patients with a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose additional risk to the patient;
* Patients with poorly controlled diabetes mellitus defined as Haemoglobin A1c level >8%;
* Patients with poorly controlled hypertension (sustained Systolic Blood Pressure of > 150 mmHg or Diastolic Blood Pressure > 95 mmHg);
* Patients with any active acute or chronic infections requiring antimicrobial therapy, or serious viral (e.g., hepatitis, herpes zoster, HIV positivity) or fungal infections;
* Patients with a history of recurrent upper gastrointestinal (UGI) ulceration or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a significant coagulation defect, or any other condition, which in the Investigator's opinion might preclude the chronic use of Celecoxib or Diacerein. Patients may, at the Investigator's discretion, take a proton pump inhibitor (PPI) or antacids daily as required, with a 2 hour period between intake of study medication and intake of PPI or antacid;
* Patients who have been diagnosed as having or have been treated for esophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to receiving the first dose of study medication;
* Patients with chronic liver or kidney disease, as defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 times the upper limit of normal (ULN) or blood urea nitrogen (BUN) or serum creatinine > 2.0 times ULN, at the Screening Visit (Visit 1);
* Patients who have a history of intolerance to acetaminophen or paracetamol, opioids or opioid combinations such that it is felt that an adequate non-anti-inflammatory rescue analgesic regimen cannot be safely prescribed;
* Patients who have a history of alcohol or substance abuse within the last 3 years;
* Patients receiving any investigational drug within 30 days or 5 half-lives (whichever is greater) prior to the Inclusion Visit (Visit 2);
* Patients who plan surgery during the study;
* Female patients who are breastfeeding;
* Patients with the impossibility of taking part in the total duration of the study and attending the visits;
* Patients unable to give an informed consent;
* Patients who do not respect the acetaminophen or paracetamol washout period of 48 hours or the NSAID washout period of 1 week before the Inclusion Visit (Visit 2).

Treatment-Related Exclusion:

* Patients using corticosteroids (oral, injectable; exception of intraarticular/soft tissue injection at the exclusion of the target knee), indomethacin, therapeutic dose of glucosamine, chondroitin sulphate or Diacerein or Avocado-Soybean Unsaponifiables (ASU) during the 12 weeks preceding inclusion (intraarticular injections of corticosteroids in the contralateral knee is allowed during the study);
* Patients using hyaluronic acid (intra-articular target knee) during the 26 weeks preceding inclusion;
* Patients using natural health products (e.g. capsaicin, boswellia, willow bark), and creams and analgesic gels (e.g. camphor and alcohol based gels) during one week preceding inclusion;
* Patients using natural health products susceptible to increase the risk of bleeding (e.g. garlic, dong quai, etc.) during one week preceding inclusion;
* Patients receiving radioactive synovectomy (target knee) during the 12 weeks preceding inclusion;
* Patients who are taking NSAIDs and do not want to stop during the study;
* If treatment of osteoporosis (bisphosphonates, selective estrogen receptor modulators [SERMS], thyroid-stimulating hormone [TSH]) is necessary, it will have to be continued, unmodified, for the entire duration of the study;
* Patients who have used compounds containing non-approved agents for arthritis or agents claiming to possess disease/structure-modifying properties in the 14 days prior to the Inclusion Visit (Visit 2);
* Patients who have used medications with matrix metalloproteinase (MMP)-inhibitory properties (e.g. tetracycline or structurally related compounds) within 28 days prior to the Inclusion Visit (Visit 2);
* Patients who require acetaminophen or paracetamol at daily doses > 2000 mg (2g) on a regular basis;
* Patients who are taking a laxative, lithium carbonate, phenytoin or anticoagulants (with the exception of ASA up to a maximum daily dose of 325 mg);
* Patients who have received chondrocyte transplants or underwent other type of cartilage repair procedures in the target joint;
* Patients who use oral or topical coxibs;
* Patients who use calcitonin;
* Patients who use immunosuppressive drugs.

Criteria-Related to Magnetic Resonance Imaging (MRI):

* Patients presenting a counter-indication to an MRI examination;
* Patients whose Inclusion Visit cartilage volume cannot be calculated from the MRI due to advanced OA disease;
* Patients whose Inclusion Visit cartilage volume cannot be calculated from the MRI due to the presence of large fat pads or any other technical reason;
* Patients with study knee not entering in the MRI magnet;
* Patients with abnormal Inclusion Visit findings and/or any other condition, which, in the Investigator's judgment, might increase the risk to the patient or decrease the chance of obtaining satisfactory data through MRI to achieve the objectives of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Pelletier, MD, FRCPC, Principal Investigator — ArthroLab Inc.; Jean-Pierre Raynauld, MD, FRCPC, Principal Investigator — Osteoarthritis Research Unit, University of Montreal Hospital Center
Locations (22):
- State Hospital Stockerau Karl Landsteiner Institute for Clinical Rheumatology, Stockerau, Austria
- Belgium (2):
  - Institut Médical Spécialisé - Centre DISCCA, Hornu
  - Reumatologie Medizorg Merksem, Merksem
- Canada (8):
  - Institut de recherche en rhumatologie de Montréal, Montreal, Quebec
  - PPS Medical Inc, Montreal, Quebec
  - Hopital du Sacré Coeur de Montréal du CIUSS du Nord-de-l'île-de-Montréal, Montreal, Quebec
  - West Island Rheumatology Research Associates, Pointe-Claire, Quebec
  - Diex Recherche Québec Inc., Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de recherche musculo-squelettique, Trois-Rivières, Quebec
  - G.R.M.O (Groupe de recherche en rhumatologie et maladies osseuses) Inc., Québec
- Czechia (4):
  - Rheumatology St. Anne's University Hospital Brno, Brno
  - Institute of Rheumatology and Clinic of Rheumatology Charles University, Prague
  - Affidea Praha, s.r.o., Prague
  - Medical Plus s.r.o., Uherské Hradiště
- Spain (7):
  - Rheumatology Hospital Universitario A Coruna, A Coruña
  - Rheumatology Instituto Poal de Reumatologia, Barcelona
  - Rheumatology Bellvitge University Hospital, Barcelona
  - Hospital Quiron, Unidad de Medicina interna, Barcelona
  - Rheumatology Hospital del Mar - Parc de Salut Mar, Barcelona
  - Universitario de Mostoles Río Júcar, Madrid
  - Departament de Reumatologia Hospital Parc Tauli de Sabadell, Sabadell

REFERENCES:
- [Background] Pavelka K, Trc T, Karpas K, Vitek P, Sedlackova M, Vlasakova V, Bohmova J, Rovensky J. The efficacy and safety of diacerein in the treatment of painful osteoarthritis of the knee: a randomized, multicenter, double-blind, placebo-controlled study with primary end points at two months after the end of a three-month treatment period. Arthritis Rheum. 2007 Dec;56(12):4055-64. doi: 10.1002/art.23056. PMID 18050202
- [Background] Bartels EM, Bliddal H, Schondorff PK, Altman RD, Zhang W, Christensen R. Symptomatic efficacy and safety of diacerein in the treatment of osteoarthritis: a meta-analysis of randomized placebo-controlled trials. Osteoarthritis Cartilage. 2010 Mar;18(3):289-96. doi: 10.1016/j.joca.2009.10.006. Epub 2009 Oct 14. PMID 19857509
- [Background] Moldovan F, Pelletier JP, Jolicoeur FC, Cloutier JM, Martel-Pelletier J. Diacerhein and rhein reduce the ICE-induced IL-1beta and IL-18 activation in human osteoarthritic cartilage. Osteoarthritis Cartilage. 2000 May;8(3):186-96. doi: 10.1053/joca.1999.0289. PMID 10806046
- [Background] Pelletier JP, Mineau F, Fernandes JC, Duval N, Martel-Pelletier J. Diacerhein and rhein reduce the interleukin 1beta stimulated inducible nitric oxide synthesis level and activity while stimulating cyclooxygenase-2 synthesis in human osteoarthritic chondrocytes. J Rheumatol. 1998 Dec;25(12):2417-24. PMID 9858439
- [Background] Martel-Pelletier J, Mineau F, Jolicoeur FC, Cloutier JM, Pelletier JP. In vitro effects of diacerhein and rhein on interleukin 1 and tumor necrosis factor-alpha systems in human osteoarthritic synovium and chondrocytes. J Rheumatol. 1998 Apr;25(4):753-62. PMID 9558181
- [Background] Franchi-Micheli S, Lavacchi L, Friedmann CA, Zilletti L. The influence of rhein on the biosynthesis of prostaglandin-like substances in-vitro. J Pharm Pharmacol. 1983 Apr;35(4):262-4. doi: 10.1111/j.2042-7158.1983.tb02929.x. No abstract available. PMID 6133942
- [Background] Petrillo M, Montrone F, Ardizzone S, Caruso I, Porro GB. Endoscopic evaluation of diacetylrhein-induced gastric-mucosal lesions. Curr Ther Res Clin Exp. 1991;49(1):10-15.
- [Derived] Pelletier JP, Raynauld JP, Dorais M, Bessette L, Dokoupilova E, Morin F, Pavelka K, Paiement P, Martel-Pelletier J; DISSCO Trial Investigator Group. An international, multicentre, double-blind, randomized study (DISSCO): effect of diacerein vs celecoxib on symptoms in knee osteoarthritis. Rheumatology (Oxford). 2020 Dec 1;59(12):3858-3868. doi: 10.1093/rheumatology/keaa072. PMID 32521015

RESULTS

PARTICIPANT FLOW:
Groups:
- Diacerein: One placebo capsule once daily in the morning (breakfast) and one diacerein 50 mg capsule once daily in the evening (dinner) for the first month, then diacerein capsules twice daily with meals in the morning (breakfast) and the evening (dinner).
  Diacerein
  Placebo
- Celecoxib: One celecoxib 200 mg capsule once daily in the morning (breakfast) and one placebo capsule once daily in the evening (dinner).
  Celecoxib
  Placebo
Period: Overall Study
Arm/Group | Diacerein | Celecoxib
Started | 187 | 193
Completed | 141 | 149
Not Completed | 46 | 44
Not completed — Protocol Violation | 2 | 5
Not completed — Lack of Efficacy | 7 | 7
Not completed — Adverse Event | 21 | 12
Not completed — Withdrawal by Subject | 15 | 13
Not completed — No study medication intake | 1 | 4
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Diacerein | Celecoxib | Total
Number analyzed (Participants) | 187 | 193 | 380
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 97 | 203
  >=65 years | 81 | 96 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (6.3) | 64.4 (7.0) | 64.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 146 | 283
  Male | 50 | 47 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 80 | 79 | 159
  Austria | 3 | 6 | 9
  Belgium | 2 | 1 | 3
  Czechia | 59 | 63 | 122
  Spain | 43 | 44 | 87
Study Knee [Number; unit: participants]
  Right knee | 87 | 96 | 183
  Left knee | 100 | 97 | 197

OUTCOME MEASURES:

1. Primary Outcome: Change Form Baseline in WOMAC A Pain Subscale
Description: Change form baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) A pain subscale after 182 days of treatment.
  WOMAC A pain subscale: 0 - 50 cm; 50 = worse
Time Frame: baseline and 182 days
Population: The Per Protocol Set (PPS) was a subset of the ITT and included all patients who did not present any major deviation of the protocol over the 6-month follow-up period. These deviations were detected during the blind review meeting.
Measure: Mean (Standard Error); unit: cm
Groups:
- Diacerein: One placebo capsule once daily in the morning (breakfast) and one diacerein 50 mg capsule once daily in the evening (dinner) for the first month, then diacerein capsules twice daily with meals in the morning (breakfast) and the evening (dinner).
  Diacerein
  Placebo
  ITT (n=
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 140 | 148
cm | -11.14 (0.91) | -11.82 (0.89)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Non-Inferiority — Non-inferiority of Diacerein versus Celecoxib was assessed by computing the difference in the adjusted mean change from baseline (Visit 2) in WOMAC Pain subscale score after 182 days of treatment between Diacerein and Celecoxib treatment groups from a MMRM. Assuming that: * Non inferiority margin of 10 points for the absolute change in WOMAC Pain Subscale Score (scale 0-100) * SD of 26 in the two treatment groups, * Type I error: α = 0.025 (one-sided condition) and power equal to 90%; p < 0.025, Mixed Models Analysis — MMRM. Non-inferiority claim:Diacerein to be non-inferior to Celecoxib if upper bound of the the difference in the adjusted mean change was inferior to 5 cm on the PPS; Mean Difference (Final Values) = 0.67, 95% CI 1-sided [upper limit 3.18]

2. Secondary Outcome: Change From Baseline in WOMAC OA Scores
Description: Absolute Changes from Baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) after 182 days of treatment.
  WOMAC scale: 0 - 240 cm; 240 = worse - Intention-To-Treat (N=370) Pain subscale: 0-50cm; 50 = worse; Stifness subscale: 0-20cm; 20 = worse; Function subscale: 0-170cm; 170 = worse Absolute changes in WOMAC scores: <0 = improvement; 0 = stable; >0 = worsening
Time Frame: Day 182 or early termination
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
score
  Total Score: number analyzed (Participants) | 177 | 182
  Total Score | -41.0 (53.1) | -42.9 (55.0)
  Pain Score: number analyzed (Participants) | 178 | 182
  Pain Score | -10.03 (11.95) | -9.60 (12.02)
  Stiffness Score: number analyzed (Participants) | 178 | 182
  Stiffness Score | -3.56 (4.99) | -3.99 (5.32)
  Physical Function Score: number analyzed (Participants) | 177 | 182
  Physical Function Score | -27.2 (39.0) | -29.3 (39.8)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Absolute Changes From Baseline in Pain Visual Analogue Scale
Description: Absolute Changes from Baseline in Pain Visual Analogue Scale (VAS): 0-10 cm; 10 = worse
Time Frame: Day 182 or early termination
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
score | -2.34 (2.55) | -2.46 (2.61)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: OARSI Responders
Description: Osteoarthritis Research Society International (OARSI) Responders
Time Frame: Day 182 or early termination
Population: Intentio-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
Participants | 99 | 97
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Chi-squared

5. Secondary Outcome: Assessment of Joint Swelling, Effusion or Both
Description: Assessment of Joint Swelling, joint Effusion or Both
Time Frame: Day 182 or early termination
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
participants
  Joint Swelling | 47 | 48
  Joint Effusion | 37 | 37
  Joint Swelling and Effusion | 19 | 23
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Chi-squared

6. Secondary Outcome: Consumption of Acetaminophen
Description: Overall Daily number of tablets taken during the 6 month study
Time Frame: Day 182 or early termination
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
tablets | 1.06 (1.75) | 0.91 (1.02)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Chi-squared

7. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity
Description: Change from baseline in global assessment of disease activity was assessed using a VAS scale (0-10cm; 10=worse)
Time Frame: Day 182 or early termination
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
score
  Patient's Global Assessment | -1.81 (2.79) | -1.97 (2.97)
  Investigator's Global Assessment | -2.02 (2.55) | -2.65 (2.55)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Global Assessment of Response to Therapy
Description: Between group comparison in Patient's and Investigator's Global Assessment of Response to Therapy using a 0-10 cm disease activity VAS scale: 0 cm = very well; 10 cm = very poorly
Time Frame: Day 182 or early termination
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
score on a scale
  Patient's Global Assessement | 3.89 (2.57) | 3.61 (2.52)
  Investigator's Global Assessment | 3.85 (2.51) | 3.35 (2.42)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Quality of Life SF-36
Description: Absolute Changes from Baseline in Physical Component Summary (PCS) and Mental Component Summary (MCS) scores from the Quality of Life questionnaire SF-36. Scale range for each component (PCS and MCS): minimum = 0, maximum = 100, with higher scores indicating better quality of life. Absolute changes in each component (PCS and MCS): >0 = improvement; 0 = stable; <0 = worsening.
Time Frame: Day 182 or early termination
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 183 | 187
score on a scale
  Physical Component Summary | 2.46 (6.74) | 4.57 (8.08)
  Mental Component Summary | 1.56 (8.34) | -0.14 (8.87)
Statistical Analysis 1: Comparison: Diacerein vs Celecoxib; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: Cartilage Volume Loss From Baseline in the Medial Compartment Using MRI
Description: Relative cartilage volume loss from baseline in the medial compartment of the knee using MRI
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: percentage of volume loss
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
percentage of volume loss | -4.8 (6.3) | -6.0 (6.7)

11. Other Pre Specified Outcome: Cartilage Volume Loss From Baseline in the Lateral Compartment Using MRI
Description: Relative cartilage volume loss from baseline in the lateral compartment of the knne using MRI
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: percentage of volume loss
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
percentage of volume loss | -4.4 (4.4) | -4.1 (4.0)

12. Other Pre Specified Outcome: Change From Baseline in Synovitis (Synovial Membrane Thickness) Using MRI
Description: Absolute Change from baseline in synovitis (synovial membrane thickness) in the global knee using MRI
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
mm | 0.24 (0.18) | 0.27 (0.15)

13. Other Pre Specified Outcome: Change From Baseline in WOMAC A Pain Subscale
Description: Relative mean change from baseline in WOMAC Pain subscore
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: percentage of change in WOMAC Pain score
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
percentage of change in WOMAC Pain score | -26.2 (48.0) | -37.1 (52.2)

14. Other Pre Specified Outcome: Change From Baseline in Global Stiffness Using WOMAC Subscale
Description: Relative Change from baseline in global stiffness using WOMAC subscale
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: percentage of change in WOMACStifness sc
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
percentage of change in WOMACStifness sc | -24.3 (46.6) | -38.1 (44.5)

15. Other Pre Specified Outcome: Change From Baseline in Visual Analogue Scale Pain (VAS-Huskisson's)
Description: Relative change from baseline in Visual Analogue Scale pain (VAS-Huskisson's)
Time Frame: baseline and 728 days
Population: Exploratory ITT
Measure: Mean (Standard Deviation); unit: Percentage of change in VAS score
Arm/Group | Diacerein | Celecoxib
Number analyzed (Participants) | 26 | 30
Percentage of change in VAS score | -31.4 (43.8) | -37.6 (44.4)

ADVERSE EVENTS:
Time Frame: At each post-screening visit up to 2 years
Description: Of the 380 randomised patients, 4 patients did not receive at least one dose of study treatment. Thus the Safety Set was composed of 376 patients: 186 (99.5%) in the Diacerein group and 190 (98.4%) in the Celecoxib group.
Arm/Group | Diacerein | Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/190
Serious Adverse Events (participants affected / at risk) | 3/186 | 4/190
Other Adverse Events (participants affected / at risk) | 49/186 | 33/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diacerein (N=186) | Celecoxib (N=190)
Temporal arteritis (Vascular disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diacerein (N=186) | Celecoxib (N=190)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chromaturia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (21) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 5 (5)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 3 (3) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematuria (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue geographic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Infections and infestations) | 2 (2) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Palpitations (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All documents, data, know-how, formulae, and unused drugs provided to the Study Site or Investigator for purposes of the Study are and will remain the sponsor's (or its agent) property.

The sponsor (or its agent) will have the right to use the results of the Study in any manner deemed appropriate to the sponsor's business interests.

The sponsor will store information regarding the Study Site and Investigator in a database system, to be used for internal sponsor assessment purposes only.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT02688400/Prot_SAP_000.pdf